CLINICAL TRIAL: NCT00003980
Title: Phase I and Pharmacokinetics Study to Determine the Safety of BIBX 1382 in Patients With a Solid Tumor on a Continuous Daily Oral Administration Schedule and After Single Oral and Intravenous Doses
Brief Title: BIBX 1382 in Treating Patients With Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16981; EORTC-16981
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: BIBX 1382

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of BIBX 1382 in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of oral BIBX 1382 in patients with solid tumors. II. Determine qualitative and quantitative toxicities of oral BIBX 1382 in these patients. III. Determine predictability, duration, intensity, onset, reversibility, and dose relationship of the toxicities of oral BIBX 1382 in these patients. IV. Determine safe and optimal doses of oral BIBX 1382 for a Phase II study. V. Assess the pharmacokinetics of oral BIBX 1382 in these patients. VI. Document any antitumor activity in these patients treated with oral BIBX 1382.

OUTLINE: This is a dose escalation study. Patients receive BIBX 1382 IV over 1 hour followed 7 days later by oral BIBX 1382. Beginning 3 days later, patients receive oral BIBX 1382 daily for 28 days. Courses of daily oral BIBX 1382 repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of oral BIBX 1382. The maximum tolerated dose (MTD) is defined as the dose at which dose limiting toxicity occurs in at least 2 of 6 patients. Patients are followed for up to 4 weeks.

PROJECTED ACCRUAL: A total of 40-80 patients will be accrued for this study over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven solid tumor not amenable to standard treatment No symptomatic brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL Other liver function tests no greater than 2 times upper limit of normal (unless related to liver metastases) Renal: Creatinine no greater than 1.4 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study No active bacterial infections No nonmalignant disease that would be incompatible with study No prior alcoholism, drug addiction, or psychotic disorders

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy (6 weeks for extensive radiotherapy) No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational or antitumor drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1999-02

CONTACTS AND LOCATIONS:
Overall Officials: Christian Dittrich, MD, Study Chair — Ludwig Boltzmann Institute for Applied Cancer Research at Kaiser Franz Josef Hospital
Locations (27):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Ludwig Institute for Cancer Research-Brussels Branch, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Herlev, Denmark
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - C.R.C. Beatson Laboratories, Glasgow, Scotland